CLINICAL TRIAL: NCT02043457
Title: Identification of Phenotypic Factors That Predict Success for Weight Loss and Long-term Weight Maintenance
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy E Rothberg, Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00030088
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Immunophenotyping; Absorptiometry, Photon; DNA; RNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA that is de-indentified is stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle intervention: Opt-in intervention to include the following procedures, called 'phenotyping' performed at baseline, after 10-15% weight loss from baseline weight or 6 months (whichever comes first) and at end of 2 years while in weight maintenance: oral glucose tolerance test, mixed meal tolerance test, with fasting leptin, biased and unbiased metabolomic profiling, DNA, RNA, muscle and adipose tissue biopsies: measurement of resting energy expenditure by indirect calorimetry; oxidative capacity (V02 peak/max); body composition by Dual Energy X-ray Absorptiometry (DEXA) or air displacement plethysmograph (Bod Pod); inventories of depression and health related quality of life instruments, measures of impulsivity, measures of hunger and appetite, work performance (including presenteeism and absenteeism) and pain survey.
  Interventions: Other: phenotyping

INTERVENTIONS:
Other: phenotyping
  Other Names: Phentoyping includes:; Health related quality of life questionnaires; Depression Inventory; Work Performance; Resting Energy Expenditure measured by indirect calorimetry; Oxidative Capacity measured by V02 max; Body composition measured by Dual Energy X-ray Absorptiometry (DEXA) or air displacement plethysmograph (Bod Pod); Mixed Meal Tolerance Testing with metabolomic profiling and hormone evaluation; Oral Glucose Tolerance Testing; DNA; RNA; Muscle biopsy (from vastus lateralis); Adipose tissue biopsy from abdomen; Survey regarding pain

SUMMARY:
The Investigational Weight Management Clinic now entitled the Weight Management Program at the University of Michigan was created to identify strategies that will result in cost-effective, long term weight management for overweight and obese individuals. The driving hypothesis of the clinic is that the 'one size fits all' philosophy is untenable with a complex disease such as obesity. The clinic will serve as a portal for patients to choose standard clinical care or to explore alternatives from a variety of clinical studies offered through the clinic. These studies will include further investigations into nutrition, the biological basis of weight and weight management and protocols using approved and experimental pharmaceuticals as well as technologies that aid in self-management of weight.

ELIGIBILITY:
Inclusion Criteria:

* Obese males and females: age >20 years; Obese population defined as BMI > or = 27 kg/m2
* Lean population BMI < 27 but > 17 kg/m2
* Able and willing to provide written informed consent for the trial

Exclusion Criteria:

* Evidence of inherited disorders of lipid metabolism.
* History of Cancer within the last 5 years
* Human immunodeficiency virus (HIV) antibody positive.
* Patients with solid organ transplants.
* Participation in any other clinical trial within 90 days of entry into this trial.
* Pregnant or lactating females.
* Uncontrolled thyroid disease
* Unstable angina or NY heart association class II failure or above
* Gastrointestinal disease specifically GI motility disorders
* Unstable neuropsychiatric disease including major depression/anxiety, eating disorder such as binge eating, bulimia or anorexia
* End stage renal or hepatic disease
* Autoimmune disorders (e.g. SLE)
* Body weight fluctuation of more than 5 kg in the previous 3 months
* Prior bariatric surgery
* A history or current alcohol/substance abuse and change in smoking habits or cessation in the past 6 months.
* Women of childbearing age must use a reliable form of contraception.
* Any medical condition, which in the opinion of the investigator would make the patient unsuitable for recruitment, or could interfere with the patient participating in or completing the protocol.
* Unwilling or unable to consent for the study.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 3000 obese participating in a 2 year clinical weight loss and weight maintenance program and 200 lean controls may opt-in to participate in a number of evaluations including depression inventory and HRQOL questionnaires, assessing hunger and appetite, work performance (including presenteeism and absenteeism), pain survey, oral glucose tolerance testing, mixed meal tolerance testing with metabolomics, DNA, RNA, with or without muscle and adipose tissue biopsies, body composition by DEXA or BodPod, measurements of REE and V02 max before at baseline, at 10-15% weight loss and after the 2 year clinical program.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2009-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phenotypic factors related to weight loss and long-term weight maintenance | Change in phenotypic factors from baseline to 3-6 months and at 2 years
  Phenotypic factors include:
  blood glucose levels, lipomic/metabolomic measurements, genetic analysis, body fat percentage, maximal oxygen consumption, respiratory quotient, resting metabolic rate, physical/emotional health

CONTACTS AND LOCATIONS:
Overall Officials: Charles Burant, MD, PhD, Study Director — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Rothberg AE, Marriott DJ, Miller NM, Herman WH. Retention and weight outcomes after transitioning an intensive behavioral weight management program from an in-person to a virtual format. Obes Sci Pract. 2023 Apr 20;9(5):452-458. doi: 10.1002/osp4.673. eCollection 2023 Oct. PMID 37810529
- [Derived] Rothberg AE, McEwen LN, Kraftson AT, Fowler CE, Herman WH. Very-low-energy diet for type 2 diabetes: an underutilized therapy? J Diabetes Complications. 2014 Jul-Aug;28(4):506-10. doi: 10.1016/j.jdiacomp.2014.03.014. Epub 2014 Mar 29. PMID 24849710
- See also: Related Info — http://www.med.umich.edu/intmed/endocrinology/weightmanagement/index.htm